CLINICAL TRIAL: NCT02971956
Title: A Phase II Study of Pembrolizumab in Refractory Advanced Esophageal Cancer
Brief Title: Pembrolizumab in Refractory Advanced Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Peter Enzinger, MD, Peter C. Enzinger MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-293
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Results first posted 2022-04-08 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Esophageal Cancer; Squamous Cell Esophagus Cancer; Adenocarcinoma Esophagus
Keywords: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Immune checkpoint inhibitor
  Other Names: Keytruda

SUMMARY:
This research study is studying a targeted therapy as a possible treatment for advanced esophageal cancer.

The study intervention involved in this study is:

-Pembrolizumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved Pembrolizumab for the participant specific disease but it has been approved for other uses.

Pembrolizumab, also known as KEYTRUDA or MK-3475, is approved in the USA and several other countries to treat other types of diseases.

The goal of this research study is to

-Evaluate the safety and efficacy of pembrolizumab in participants with advanced esophageal cancer that have not responded to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, measurable, unresectable adenocarcinoma or squamous cell carcinoma of the esophagus. For the purposes of this study, undifferentiated carcinomas or adenosquamous carcinomas will be categorized as adenocarcinomas.
* The primary tumor must originate in the esophagus. Tumors that involve the GE junction must meet Sievert Type 1 criteria: "Adenocarcinoma of the distal oesophagus which usually arises from an area with specialized intestinal metaplasia of the oesophagus (i.e. Barrett's oesophagus) and which may infiltrate the oesophagogastric junction from above." For the purposes of this protocol, this will be interpreted as: greater than 50% of the tumor must be above the GE junction or, alternatively, the tumor must involve the GE junction and arise in the setting of biopsy-documented Barrett's esophagus (specialized intestinal metaplasia).
* Patients must have received at least one prior therapy for unresectable disease. Patients with recurrence within 6 months of completion of neoadjuvant or adjuvant therapy may be considered as having received one prior therapy for unresectable disease.
* Be willing and able to provide written informed consent/assent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Have measurable disease based on irRECIST.
* Be willing to provide tissue from a newly obtained biopsy of a tumor lesion, most commonly an EGD biopsy from the esophagus. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor. Please note, patients may not initiate therapy until the biopsy specimen is received at the Dana-Farber Cancer Institute.
* The first 15 patients with adenocarcinoma will be offered an optional tumor biopsy (typically EGD biopsy) at 8 weeks. Starting with adenocarcinoma patient #16, patients must have an accessible tumor and must agree to tumor biopsy at 8 weeks; this will continue to be mandatory until a total of 20 patients have undergone biopsy at 8 weeks.
* Have a performance status of 0 or 1 on the ECOG Performance Scale (Appendix A).
* Female subject of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 6.3.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Demonstrate adequate organ function as defined below, all screening labs should be performed within 10 days of treatment initiation.

Hematological

* Absolute neutrophil count (ANC) ≥1,500 /mcL
* Platelets ≥80,000 / mcL
* Hemoglobin ≥8.5 g/dL or ≥5.6 mmol/L

  -Renal
* Serum creatinine ≤1.5 X upper limit of normal (ULN) OR Measured creatinine clearance ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (GFR can also be used in place of creatinine or CrCL) Creatinine clearance should be calculated per institutional standard.

  -Hepatic
* Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* AST (SGOT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
* ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
* Albumin > 2.8 mg/dL

  -Coagulation
* International Normalized Ratio (INR) OR Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Subjects requiring systemic steroids are excluded from the trial. The use of physiologic doses of corticosteroids may be approved after discussion with the sponsor.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with ≤ Grade 2 neuropathy and alopecia are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, they must wait ≥ 3 weeks prior to starting study treatment. They must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has an active infection requiring systemic therapy.
* Patients that require supplemental oxygen are excluded.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

  --Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2020-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C. Enzinger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: from January 2017 to October 2018
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 49
Age, Customized [Median (Full Range); unit: years] | 64 [34 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 44
  Black or African American | 2
  Asian | 1
  Other | 1
  More than one race | 1
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was evaluated each cycle on treatment; Treatment continued until disease progression or unacceptable toxicity. Treatment duration was a median of 2.1 months with a maximum of 14.9 months.
Measure: Number (95% Confidence Interval); unit: proportion of participant
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 49
proportion of participant | 0.08 [0.023 to 0.196]

2. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated each cycle on treatment and in long-term follow-up every 12 weeks for up to 5 years. Maximum follow-up in this study cohort was 28.9 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 49
months | 1.8 [1.8 to 2.0]

3. Secondary Outcome: Median Overall Survival (OS)
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: Disease was evaluated each cycle on treatment and in long-term follow-up every 12 weeks for up to 5 years. Maximum follow-up in this study cohort was 38.7 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 49
months | 5.8 [4.0 to 9.5]

4. Secondary Outcome: Number of Patients Experiencing Grade 3-4 Treatment-Related Toxicity
Description: All grade 3-4 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4 as reported on case report forms were counted. Outcome defined as the number of patients experiencing at least one treatment-related grade 3-4 AE of any type during the time of observation.
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment. Median treatment duration for this study cohort was 2.1 months with maximum of 14.9 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 49
Participants | 6

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment. Median treatment duration for this study cohort was 2.1 months with maximum of 14.9 months. All-Cause Mortality was evaluated each cycle on treatment and in long-term follow-up every 12 weeks for up to 5 years. Maximum follow-up in this study cohort was 38.7 months.
Description: Serious adverse events (AEs) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. All remaining events regardless of treatment attribution were classified as Other AEs. Maximum grade toxicity by type for a patient over time was calculated. No further data is available to specify classification of other beyond the general term.
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 49/49
Serious Adverse Events (participants affected / at risk) | 6/49
Other Adverse Events (participants affected / at risk) | 46/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=49)
Cardiac arrest (Cardiac disorders) | 1
Eye disorders - Other (Eye disorders) | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nervous system disorders - Other (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=49)
Anemia (Blood and lymphatic system disorders) | 32
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Chest pain - cardiac (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 8
Endocrine disorders - Other (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Eye disorders - Other (Eye disorders) | 2
Vitreous hemorrhage (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 15
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 17
Diarrhea (Gastrointestinal disorders) | 14
Dry mouth (Gastrointestinal disorders) | 3
Duodenal hemorrhage (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 18
Esophageal hemorrhage (Gastrointestinal disorders) | 2
Esophageal pain (Gastrointestinal disorders) | 1
Esophageal perforation (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3
Gastrointestinal pain (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 20
Obstruction gastric (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 12
Death NOS (General disorders) | 3
Edema limbs (General disorders) | 7
Fatigue (General disorders) | 40
Fever (General disorders) | 3
Gait disturbance (General disorders) | 1
General disorders and administration site conditions - Other (General disorders) | 3
Localized edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 4
Pain (General disorders) | 7
Abdominal infection (Infections and infestations) | 1
Bronchial infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 26
Aspartate aminotransferase increased (Investigations) | 20
Blood bilirubin increased (Investigations) | 7
Creatinine increased (Investigations) | 3
Investigations - Other (Investigations) | 2
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 12
Weight gain (Investigations) | 1
Weight loss (Investigations) | 10
White blood cell decreased (Investigations) | 4
Acidosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 21
Dehydration (Metabolism and nutrition disorders) | 8
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 31
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 31
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 16
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Ataxia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 2
Nervous system disorders - Other (Nervous system disorders) | 5
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 10
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 4
Confusion (Psychiatric disorders) | 7
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 6
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Renal and urinary disorders - Other (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 21
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 3
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 29
Hypotension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 3
Vascular disorders - Other (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT02971956/Prot_SAP_000.pdf